CLINICAL TRIAL: NCT01378169
Title: Early Detection and Diagnostic Performance of Bio-markers During Bacterial Sepsis: Multicentre Cohort Study in Intensive Care
Brief Title: SIRS and Bacterial Sepsis Discrimination by Biomarkers in ICU
Acronym: Captain
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: BioMérieux (Industry); Institut Pasteur (Industry); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM09143; N° 2010-A00908-31 (Other: AFSSAPS)
Record Dates: First submitted 2011-05-09; First posted 2011-06-22 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-03

CONDITIONS: SIRS; Sepsis; Severe Sepsis; Septic Shock
Keywords: SIRS; Sepsis; Severe Sepsis; Septic Shock; Inflammatory processes; Cytokines; HLA-DR; HLA type II; Chemokines; TLR expression; mRNA expression in whole blood; Bacterial DNA detection; Prognosis factors; Infection; Diagnosis
MeSH Terms: conditions — Sepsis; Shock, Septic; Infections; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, urin, CSF, BAL
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SIRS patients: Every patient, without exclusion criteria, presenting with SIRS during an hospitalization in ICU.

SUMMARY:
Aim of the study : The primary aim of the investigators study is to highlight the presence of biomarkers (biological indicators of the presence of inflammation or infection) of infectious processes during the systemic inflammatory response (SIRS) allowing, first to discriminate non-infectious inflammation from infectious processes and secondary to determine the microbial pathogen responsive of the infection. For this purpose the investigators will conduct a combinatorial approach of several blood markers including usual markers of inflammation and other blood and cells markers. Expression of small pieces of RNA (miRNA) known to inhibit determined gene expression, will also be analysed in monocytes (a specific group of white blood cells involved in the fist line of defences against microbes.

Study design : For this purpose the investigators will include 300 patients admitted to the intensive care unit with suspicion of infection. Serial blood sample will be take for biological parameters analysis. Efficiency of each single parameters and of different combinations of different markers to determine the presence or absence of infection responsive of clinical inflammation will be studied.

DETAILED DESCRIPTION:
Aim of the study : The project's main objective is the establishment of the diagnostic performance of the association of diagnostic markers of infectious processes linked to the pathogen or host during the systemic inflammatory response syndromes (SIRS) in critical care patients allowing, first to discriminate non infectious SIRS from sepsis and, secondary to determine the microbial pathogen responsive of the inflammation. For this purpose, we will conduct a combinatorial approach of several plasma markers including usual markers (CRP, PCT, other soluble mediators (soluble TREM-1, IL-6, IL-1Ra, IL-10, CXCL2, CXCL8, CCL2 and CCL5), cell markers (CD14 / HLA-DR expression on monocytes and TLR2, 4, 9 expression on NK cells) together with modified expression of microRNA (miRNA) in circulating monocytes.

Study design : This study will include patients admitted to the ICU with SIRS and suspected sepsis, according to usual criteria. Infection definition will be based on a combination clinical, bacteriological and cyto-or histo-pathological according to the disease involved.

A serial measurement of biological parameters previously described will be realized from D0 to D3.

Evaluation criteria : The primary endpoint is to determine the ability of each individual parameter and of the different combination to discriminate between sepsis and noninfectious inflammation. The diagnostic performance of biomarkers studied will be done by calculating the sensitivity, specificity, positive and negative predictive value of each test alone or in combination with respect to the existence of an infection (sepsis) or not (SIRS). According to data from the literature and our own experience, the expected proportion of patients with sepsis among the holders of SIRS was 50%. The discriminatory ability of each test will be performed by using ROC curves and calibration using the Hosmer-Lemeshow several layers of increasing severity. The level of service provided is a p-value <5%. There are no plans to statistical criteria for stopping the search in case of biological data missing.

The value of the area under the ROC curve (AUC) of the PCT is 78% (95% CI 69-77). Assuming that one of the tests or combinatorial approach will increase the AUC to 85%, the number of patients needed for this study is estimated to be 300.

Conduct of research : Study will be conducted in 5 different sites. Patients admitted with or who develop a SIRS during hospitalization will be included. There will be nothing peculiar in the therapeutic management and patients will be covert by the international guidelines.

* Inclusion criteria:

  * Patient admitted with or who develop SIRS during ICU hospitalisation
  * Two or more parameter of the SIRS definition
  * Patient does not preclude its participation in the study
* Non inclusion criteria

  * Decision of withdrawal or withholding therapeutic interventions
  * No affiliation to a social security scheme

The measurement of biological endpoints will be conducted once daily, from D0 (admission) to D2 using a blood sample. The study of monocyte expression of miRNA will be performed on a portion of the cohort, corresponding to patients selected on the St. Joseph site (intensive care unit and surgical intensive care unit) because of complexity to implement, and cost level (requiring specific funding).

Total projected duration of the search: The recruitment period will run for 23 months with the aim to include all 300 patients. Patients included in the research will be followed until day 28 or day of hospital leaving, if earlier.

Stopping rules of the study to a patient: patient can discontinue their participation at any time during the research.

Security evaluation : Being a non-interventional study (biological collection) in the usual care of patients, no serious adverse event is expected to be related to research.

Any new data security, potentially leading to a reassessment of the benefits and risks of research, or which may be sufficient to consider changes in the conduct of research must be reported.

ELIGIBILITY:
Inclusion Criteria:

* Age> = 18 years
* Patient hospitalized in ICU with a diagnosis of SIRS:
* Temperatures above 38 ° C or below 36 ° C

At least one other criterion from:

* Heart rate> 90 bpm
* Respiratory rate above 20 breaths / min or PaCO2 <32 mmHg
* Leukocytosis greater than or less than 4000/mm3 12000/m3

  * Patient admitted in intensive care for less than 12 hours
  * Patient does not preclude its participation in the study.

Exclusion Criteria:

* Decision to limit treatment before potential inclusion in the study
* No affiliation to a social security scheme (beneficiary or assignee)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients whatever was their admission indication presenting a SIRS with or without sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2013-06-01 (Actual)

PRIMARY OUTCOMES:
Combination of biomarkers in sepsis | 3 days ( from D0 to D2)
  The primary endpoint is to determine the ability of each individual parameter and of the different combination to discriminate between sepsis and noninfectious inflammation.
  Each biomarker will be isolatelly studied to determine existence of a cut-off value allowing discrimination between SIRS and sepsis.
  Each positive biomarker (biomarker for which such a cut-off can be determined), will be include in a second study involving all or part of the positive biomarkers to determine the possibility of increasing AUC for discrimination of SIRS and sepsis patients

SECONDARY OUTCOMES:
Pathogen in human fluids (Blood, BAL, CSF, Urin) | D0
  A partnership with Biomerieux laboratory was estabished to allow microbial detection at D0 by a new system of microbial DNA amplification, which is at the moment under development
mRNA expression during inflammatory process in white blood cells | D0 to D3
  Study of modification of mRNA expression between SIRS and sepsis during inflammatory process in white blood cells. Study of the expression of whole mRNA in whole blood and of its modification during the 3 fist days of SIRS to determine a potential specific profil during infectious processes

CONTACTS AND LOCATIONS:
Overall Officials: François J Philippart, MD; PhD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe hospitalier Paris Saint Joseph, Paris, France

REFERENCES:
- [Background] Annane D, Bellissant E, Cavaillon JM. Septic shock. Lancet. 2005 Jan 1-7;365(9453):63-78. doi: 10.1016/S0140-6736(04)17667-8. PMID 15639681
- [Background] Gibot S, Cravoisy A, Levy B, Bene MC, Faure G, Bollaert PE. Soluble triggering receptor expressed on myeloid cells and the diagnosis of pneumonia. N Engl J Med. 2004 Jan 29;350(5):451-8. doi: 10.1056/NEJMoa031544. PMID 14749453
- [Background] Adib-Conquy M, Monchi M, Goulenok C, Laurent I, Thuong M, Cavaillon JM, Adrie C. Increased plasma levels of soluble triggering receptor expressed on myeloid cells 1 and procalcitonin after cardiac surgery and cardiac arrest without infection. Shock. 2007 Oct;28(4):406-10. doi: 10.1097/shk.0b013e3180488154. PMID 17558349
- [Background] Cavaillon JM, Adib-Conquy M, Fitting C, Adrie C, Payen D. Cytokine cascade in sepsis. Scand J Infect Dis. 2003;35(9):535-44. doi: 10.1080/00365540310015935. PMID 14620132
- [Background] Adrie C, Adib-Conquy M, Laurent I, Monchi M, Vinsonneau C, Fitting C, Fraisse F, Dinh-Xuan AT, Carli P, Spaulding C, Dhainaut JF, Cavaillon JM. Successful cardiopulmonary resuscitation after cardiac arrest as a "sepsis-like" syndrome. Circulation. 2002 Jul 30;106(5):562-8. doi: 10.1161/01.cir.0000023891.80661.ad. PMID 12147537
- [Background] Monneret G, Lepape A, Voirin N, Bohe J, Venet F, Debard AL, Thizy H, Bienvenu J, Gueyffier F, Vanhems P. Persisting low monocyte human leukocyte antigen-DR expression predicts mortality in septic shock. Intensive Care Med. 2006 Aug;32(8):1175-83. doi: 10.1007/s00134-006-0204-8. Epub 2006 Jun 2. PMID 16741700
- [Background] Munoz C, Carlet J, Fitting C, Misset B, Bleriot JP, Cavaillon JM. Dysregulation of in vitro cytokine production by monocytes during sepsis. J Clin Invest. 1991 Nov;88(5):1747-54. doi: 10.1172/JCI115493. PMID 1939659
- [Derived] Misset B, Philippart F, Fitting C, Bedos JP, Diehl JL, Hamzaoui O, Annane D, Journois D, Parlato M, Moucadel V, Cavaillon JM, Coste J; CAPTAIN Study Group. Clustering ICU patients with sepsis based on the patterns of their circulating biomarkers: A secondary analysis of the CAPTAIN prospective multicenter cohort study. PLoS One. 2022 Oct 27;17(10):e0267517. doi: 10.1371/journal.pone.0267517. eCollection 2022. PMID 36301921